CLINICAL TRIAL: NCT01383577
Title: Double-blind Randomized Controlled Study of Single Versus Triple Rubber Band Ligation of Hemorrhoids
Brief Title: Comparison Between Single and Triple Rubber Band Ligation for the Treatment of Hemorrhoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Amazonas (Other)
Responsible Party: Principal Investigator, Ivan Tramujas da Costa e Silva, PhD, Federal University of Amazonas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP-S/0001/2010
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Second-degree Hemorrhoids
Keywords: Hemorrhoids; Ligation; Pain; Morbidity; Patient Satisfaction; Cost-Benefit Analysis
MeSH Terms: conditions — Hemorrhoids; Pain; Patient Satisfaction | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single hemorrhoidal ligation (Experimental): Effective ligation of one hemorrhoidal group and sham ligation of the two other major hemorrhoidal groups is performed in each session of treatment.
  Interventions: Procedure: Single hemorrhoidal ligation
- Triple hemorrhoidal ligation (Experimental): The three major hemorrhoidal groups are ligated in the first session of ligation. The three following monthly appointments of patients of this arm are for sham hemorrhoidal ligations and final revision.
  Interventions: Procedure: Triple hemorrhoidal ligation

INTERVENTIONS:
Procedure: Single hemorrhoidal ligation — Effective ligation of one hemorrhoidal group and sham ligation of the two other major hemorrhoidal groups is performed in each of three sessions of treatment. Final revision is performed 90 days after first session of hemorrhoidal ligation.
  Other Names: Rubber band ligation of hemorrhoids, single
  Arms: Single hemorrhoidal ligation
Procedure: Triple hemorrhoidal ligation — The three major hemorrhoidal groups are ligated in the first session of ligation. Sham triple hemorrhoidal ligations are performed 30 and 60 days after the first session. Final revision is done 90 days after first ligation session.
  Other Names: Rubber band ligation of hemorrhoids, multiple
  Arms: Triple hemorrhoidal ligation

SUMMARY:
Rubber band ligation is a widely adopted treatment of internal hemorrhoids in busy coloproctology institutions. All three major hemorrhoidal clusters (left lateral, right anterior and right posterior) use to be ligated in order to obtain therapeutic success. It is commonly performed either through the ligation of a single hemorrhoid per session spaced by some few weeks to the second and third sessions, or of all three major hemorrhoids in one single session. Advocates of either method of hemorrhoidal ligation have arguments to defend their choice in terms of advantages, supported mainly on personal preferences. The investigators objective is to determine, through a controlled double-blinded randomized study, if there is any superiority of single hemorrhoidal ligation per session (in a total of three sessions) over the method of ligation of all three main hemorrhoids in a sole session in terms of therapeutic success (resolution of pre-ligation symptoms), morbidity, patient satisfaction and costs (institutional, labor and patient-related).

DETAILED DESCRIPTION:
Because of conflicting results in existing literature in relation to features such as pain and immediate effectiveness of single or multiple rubber band ligation of hemorrhoids and because in the literature consulted no study was found that addressed economical features comparing single with multiple rubber band ligation of hemorrhoids, this study was designed to compare, in a double blinded, randomized and controlled model, the results of single hemorrhoidal ligation in three sessions with triple hemorrhoidal in a sole session in terms of immediate effectiveness, patient satisfaction and costs.

Patients enrolled in the study, after applying inclusion and exclusion criteria, signed the consent form, and responded to a questionaire about epidemiological data and hemorrhoidal symptoms, are (and will be) randomly allocated to one of the two arms of the study: G1: a single major hemorrhoidal group is ligated in each of three sessions of hemorrhoidal ligation, while the two other hemorrhoidal groups are submitted to sham ligation (a McGown aspirating type of hemorrhoidal ligator is employed); G2: all three major hemorrhoidal groups are ligated in the first session of treatment and in the next two sessions only sham ligations are performed. Three sessions of hemorrhoidal and/or sham ligation are performed in all patients, each spaced by one month from the other. A final consultation is held 1 month after the third ligation session in order to gather all the results of the treatment.

After each session of hemorrhoidal ligation patients receive a chart containing a modified level of pain scale (Wong & Baker) and are asked to indicate pain level (from 0 to 5: 0 = no pain, 5 = unbearable pain) at fixed intervals (immediate post-ligation, 12 h post-ligation, 24 h post-ligation and each other day until 7 days post-ligation). Investigators gather this information about pain, and patient well-being post-ligations, from 8 programmed telephone calls to the patients after each session of hemorrhoidal (or sham) ligation.

Three months after the first session of hemorrhoidal ligation all patients are examined in order to observe treatment effectiveness and gather data about complications, patient satisfaction, number of days of occupational absenteeism linked to each session of treatment and number of analgesic pills necessary for pain relief.

Comparative costs of each modality of ligation are raised taking into consideration the salaries of health professionals involved in the treatment, the salaries of the patients (calculation of absenteeism), the value of consumables used in each session of effective ligation, the depreciation price of permanent material employed and the price of medications patients have to buy.

Patients are blinded to the modality of hemorrhoidal ligation employed and the statistician does not know the nature of each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with second-degree hemorrhoids

Exclusion Criteria:

* Patients with special needs
* Immunodepression
* Indians
* Infectious, inflammatory or tumoral anorectal comorbidities
* Previous anorectal surgeries
* Patients on anticoagulant therapy or with coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Ligature-related pain intensity | 7 days
  Patients are asked to record pain intensity related to the hemorrhoidal ligation performed in a chart containing a modified pain intensity visual scale (Wong & Baker). Investigators inquire patients about immediate pain sensation after a ligation session and at regular intervals, by telephone calls, until the 7th post-treatment day (12 h, 24 h, 2nd day, 3rd day, 4th day, 5th day, 6th day and 7th day).

SECONDARY OUTCOMES:
Immediate complications | 30 days
  Complications eventually ocurring until 30 days of each session of rubber band ligation of hemorrhoids (effective or sham) are recorded by the investigators.
Resolutive capacity of rubber band ligation of hemorrhoids | 90 days
  Resolution of pre-ligation hemorrhoidal symptoms is investigated 3 months after first session of rubber band ligation of hemorrhoids.
Degree of patient satisfaction | 90 days
  Three months after first session (or single session, according to the arm of treatment) of rubber band hemorrhoidal ligation each patient degree of satisfaction with the method is recorded analogously using the modified visual pain scale of Wong & Baker.
Costs of each of the modes of ligation | 90 days
  Three months after the first rubber band ligation session, the costs involved in each treatment modality is raised. Calculations are done taking into account the value of the material employed in all the ligation sessions that are necessary to treat each individual patient, the value of the fraction of the investigators' salaries compromised in the treatment of each individual patient, how much each patient spends in pain medication and the value of the fraction of the patients' salaries involved in occupational absenteeism.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan T Costa e Silva, PhD, Principal Investigator — Universidade Federal do Amazonas; Érico L Melo, Med Grad, Study Chair — Universidade Federal do Amazonas; Giselle L Afonso, Med Grad, Study Chair — Universidade Federal do Amazonas; Felicidad S Gimenez, MSc, Study Chair — Universidade Federal do Amazonas; Shymmene O Cardoso, BAccount, Study Chair — Universidade Federal do Amazonas; Daniel Richard M Mota, Med Grad, Study Chair — Universidade Federal do Amazonas; Rachel M Carvalho, Med Grad, Study Chair — Universidade Federal do Amazonas; Saskia Regina F Coppens, Med Grad, Study Chair — Universidade Federal do Amazonas; Themis C Abensur, MSc, Study Chair — Federal University of Amazonas
Locations (1):
- Hospital Universitário Getúlio Vargas - Ambulatório Araújo Lima, Manaus, Amazonas, Brazil